CLINICAL TRIAL: NCT00349687
Title: Practicing Self-Control Lowers the Risk of Smoking Lapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Albany (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Muraven, Associate Professor, University at Albany
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DA016131; R01DA016131 (NIH)
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Behavior, Addictive; Cigarette Smoking
MeSH Terms: conditions — Behavior, Addictive; Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: self-control practice

SUMMARY:
The proposed study will investigate the role of self-control in smoking cessation and whether interventions that improve self-control can help reduce the risk of lapsing among smokers who wish to quit. Our model predicts that the regular practice of self-control should lead to a building of strength and a general improvement in self-control performance. Hence, smokers who practice self-control prior to quitting should be more likely to succeed in their cessation attempt than smokers who do not practice self-control

ELIGIBILITY:
Inclusion Criteria:

* smoked at least 10 cigarettes per day for at least two years
* currently smoking

Exclusion Criteria:

* have at least an 8th grade education level
* have a working touch-tone phone
* report low motivation and efficacy to quit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2004-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
smoking cesssation | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mark Muraven, Ph.D., Principal Investigator — University at Albany
Locations (1):
- University at Albany, Albany, New York, United States